CLINICAL TRIAL: NCT05582486
Title: Effectiveness of the Education Program for Preventing Obstetric Violence to mi̇dwi̇fe and Nurses:Results of Ebe, Nurses and Women Taking Care
Brief Title: The Effectiveness of The Training Program Given to Midwives and Nurses to Prevent Obstetric Violence
Acronym: Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, nurten özçalkap, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-1235
Record Dates: First submitted 2022-05-19; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Counseling
Keywords: obstetric violence; communication; care; midwife; nurse
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obstetric violence prevention education intervention (Experimental): The training program for the prevention of obstetric violence was given to the midwives and nurses in the experimental group by the researcher in the form of group training in the training hall of the relevant institution. The trainings were completed in a total of 16 sessions, two sessions a day and four sessions a week. Sessions were held between 16:00 and 18:00 on weekdays, each lasting approximately 40-45 minutes, with a 10-minute break between sessions. Thus, the training program applied to the experimental group was completed in 4 weeks.
  The main purpose of the training program is to prevent obstetric violence perpetrated by midwives and nurses. The training content created for this purpose included the definition of obstetric violence, pregnant and fetus rights, factors causing obstetric violence and strategies to be used to reduce obstetric violence.
  Other Names:
  • group-ED
  Interventions: Behavioral: obstetric violence prevention education intervention
- Standard of care (Experimental): Midwives and nurses in this group did not perform any practice.
  . group- SB
  Interventions: Behavioral: obstetric violence prevention education intervention

INTERVENTIONS:
Behavioral: obstetric violence prevention education intervention — While the training program for the prevention of obstetric violence consisting of 16 sessions was applied by the researcher to the midwives and nurses in the experimental group, no intervention was applied to the midwives and nurses in the control group.

SUMMARY:
In the study, 84 midwives and nurses working in hospital delivery and puerperal services and family health centers in Adiyaman province constituted the experimental group, and the control group of 84 midwives and nurses working in the delivery room and postpartum services of hospital Child and Gynecology Hospital in Malatya and family health centers', determined by randomization in the study. While the training program for the prevention of obstetric violence consisting of 16 sessions was applied by the researcher to the midwives and nurses in the experimental group, no intervention was applied to the midwives and nurses in the control group. The second phase of the study was conducted with women who received care from the hospital delivery and postpartum services and family health centers in Adiyaman province before and after the training program applied to the midwives and nurses in the experimental group (158 women before the training, 158 after the training). Data were collected with Introductory Information Forms, Caring Behaviors Inventory-30, Communication Skills Scale and Care Satisfaction Evaluation Form.

DETAILED DESCRIPTION:
The research was conducted between November 2020 and December 2021. In the study, 84 midwives and nurses working in hospital delivery and puerperal services and family health centers in Adiyaman province constituted the experimental group, and the control group of 84 midwives and nurses working in the delivery room and postpartum services of hospital Child and Gynecology Hospital in Malatya and family health centers', determined by randomization in the study. While the training program for the prevention of obstetric violence consisting of 16 sessions was applied by the researcher to the midwives and nurses in the experimental group, no intervention was applied to the midwives and nurses in the control group. The second phase of the study was conducted with women who received care from the hospital delivery and postpartum services and family health centers in Adiyaman province before and after the training program applied to the midwives and nurses in the experimental group (158 women before the training, 158 after the training). Data were collected with Introductory Information Forms, Caring Behaviors Inventory-30, Communication Skills Scale and Care Satisfaction Evaluation Form.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Those who do not have any problems during pregnancy, birth and postpartum period (such as heart disease, preeclampsia, diabetes, difficult birth, fetal anomaly),
* No psychological health problems according to medical records,
* Those who are open to communication and cooperation.

Exclusion Criteria:

* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Caring Behaviors Scale-30 | through study completion, an average of 1 year
  Caring Behaviors Inventory-30: Wolf et al. In 1994, he evaluated patient care from a philosophical and ethical point of view (136). The scale consists of 30 items and consists of three sub-dimensions: respect for others, professional knowledge and attitude, and accessibility by the individual. The 6 Likert-type scales have options never (1), rarely (2), sometimes (3), usually (4), almost always (5), and always (6). The minimum score that can be obtained from the total of the scale is 30, and the maximum score is 180. The minimum score that can be obtained from each sub-dimension of the scale is 10, and the maximum score is 60. As the sub-dimension and total scale score increase, the care perception of patients and/or caregivers increases positively.
Communication Skills Scale | through study completion, an average of 1 year
  It was developed by Korkut in order to understand how individuals evaluate their communication skills. The scale, which is a five-point Likert type, consists of 25 statements. The scale has options never (0), rarely (1), sometimes (2), often (3), and always (4). The minimum score that can be obtained from the scale is 0, and the maximum score is 100. As the scores obtained from the scale increase, it means that individuals evaluate their communication skills positively. The Cronbach's alpha reliability coefficient of the scale was found to be 0.80. In this study, α=0.94 of the scale was found.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten ÖZÇALKAP, Msc, Principal Investigator — Adiyaman Training and Research Hospital
Locations (1):
- İnönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data may be obtained either from study investigators.

REFERENCES:
- [Background] Mannava P, Durrant K, Fisher J, Chersich M, Luchters S. Attitudes and behaviours of maternal health care providers in interactions with clients: a systematic review. Global Health. 2015 Aug 15;11:36. doi: 10.1186/s12992-015-0117-9. PMID 26276053
- See also: Manuscript full text — https://globalizationandhealth.biomedcentral.com/track/pdf/10.1186/s12992-015-0117-9.pdf